CLINICAL TRIAL: NCT01461369
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose, Parallel-Group, Efficacy and Safety Study of Diclofenac [Test] Capsules in Subjects With Osteoarthritis of the Knee or Hip
Brief Title: Study of Diclofenac Capsules to Treat Osteoarthritis Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIC3-08-05
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Capsules 35 mg bid (Experimental)
  Interventions: Drug: Diclofenac
- Diclofenac Capsules 35 mg tid (Experimental)
  Interventions: Drug: Diclofenac
- Placebo Capsule (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac — 35 mg bid Capsules
  Arms: Diclofenac Capsules 35 mg bid
Drug: Diclofenac — 35 mg tid Capsules
  Arms: Diclofenac Capsules 35 mg tid
Drug: Placebo — Capsules
  Arms: Placebo Capsule

SUMMARY:
The purpose of this study is to determine whether Diclofenac [Test] Capsules are safe and effective for the treatment of osteoarthritis pain of the hip or knee.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Functional Class I-III OA of the hip or knee with documented osteoarthritis flare at baseline
* Chronic user of nonsteroidal anti-inflammatory drugs (NSAIDs) and/or acetaminophen for OA pain
* Discontinued all analgesic therapy at Screening
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control

Exclusion Criteria:

* History of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, or any NSAIDS, including diclofenac
* Requires continuous use of opioid or opioid combination products to control OA pain of the knee or hip
* Clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease
* Significant difficulties swallowing capsules or unable to tolerate oral medication
* Previous participation in another clinical study of Diclofenac Capsules or received any investigational drug or device or investigational therapy within 30 days before Screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Agaiby, MD, Principal Investigator — Clinical Investigation Specialists, Inc; Eddie Armas, MD, Principal Investigator — Well Pharma Medical Research, Corporation; Matthew Barton, MD, Principal Investigator — Office of Matthew Barton, MD; David Bouda, MD, Principal Investigator — Heartland Clinical Research, Inc; Venkata Challa, MD, Principal Investigator — Peters Medical Research; John Champlin, MD, Principal Investigator — Med Center; Francisco Chevres, MD, Principal Investigator — Pinnacle Trials, Inc; Melanie Christina, MD, Principal Investigator — Clinical Investigations of Texas, LLC; James R Clark, MD, Principal Investigator — Charlottesville Medical Research Center, LLC; Stephen Daniels, DO, Principal Investigator — Premier Research Group - Austin; Richard R Eckert, MD, Principal Investigator — Hypothetest, LLC; Brandon Essink, MD, Principal Investigator — Meridian Clinical Research; Richard M Glover, MD, Principal Investigator — Heartland Research Associates, LLC; Kent S Hoffman, DO, Principal Investigator — Alliance Clinical Research; Curtis S Horn, MD, Principal Investigator — Quality Research Inc; Raymond E Jackson, MD, Principal Investigator — Quest Research Institute; Jeffry Jacqmein, MD, Principal Investigator — Jacksonville Center For Clinical Research; Enrico Jones, MD, Principal Investigator — Triad Clinical Research; Alan Kivitz, MD, Principal Investigator — Altoona Center for Clinical Research; Kevin Kuettel, MD, Principal Investigator — ACRI-Phase I, LLC; Gregory F Lakin, DO, Principal Investigator — Professional Research Network of Kansas, LLC; Theresia Lee, MD, Principal Investigator — Progressive Clinical Research; Sathish Modugu, MD, Principal Investigator — Drug Trials America; Julie A Mullen, DO, Principal Investigator — Sterling Research Group, Ltd; Kashyap Patel, MD, Principal Investigator — Peninsula Research, Inc; Kyle Patrick, DO, Principal Investigator — Premier Research Group - Phoenix; Antoinette A Pragalos, MD, Principal Investigator — Community Research; Larry D Reed, MD, PhD, Principal Investigator — Healthcare Research; Eli M Roth, MD, Principal Investigator — Sterling Research Group, Ltd; Douglas R Schumacher, MD, Principal Investigator — Radiant Research, Inc; Mark Stich, DO, Principal Investigator — Westside Center for Clinical Research; Bradley Swenson, MD, Principal Investigator — Radiant Research, Inc; Marvin Tark, MD, Principal Investigator — Drug Studies America; Gary Tarshis, MD, Principal Investigator — Expresscare Clinical Research; Haydn M Thomas, MD, Principal Investigator — Clinical Trials Technology Inc; Cindy Tuten, MD, Principal Investigator — Clinical Study Center of Asheville, LLC; Larkin T Wadsworth, MD, Principal Investigator — Sundance Clinical Research, LLC; Robert J Wagner, MD, Principal Investigator — Community Research; Larry S Watkins, MD, Principal Investigator — Lynn Institute of the Ozarks; Tamela Zimmerman, MD, Principal Investigator — Community Research
Locations (38):
- United States (38):
  - Premier Research Group - Phoenix, Phoenix, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Acri-Phase I, LLC, Anaheim, California
  - Med Center, Carmichael, California
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Well Pharma Medical Research, Corporation, Miami, Florida
  - Peninsula Research, Inc, Ormond Beach, Florida
  - Alliance Clinical Research, Winter Park, Florida
  - Pinnacle Trials, Inc, Atlanta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Heartland Research Associates, LLC, Newton, Kansas
  - Clinical Trials Technology Inc, Prairie Village, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Quest Research Institute, Bingham Farms, Michigan
  - Healthcare Research, Florissant, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Office of Matthew Barton, MD, Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Triad Clinical Research, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Radiant Research, Inc, Columbus, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Radiant Research, Inc, Anderson, South Carolina
  - Premier Research Group - Austin, Austin, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Hypothetest, LLC, Roanoke, Virginia

REFERENCES:
- [Derived] Gibofsky A, Hochberg MC, Jaros MJ, Young CL. Efficacy and safety of low-dose submicron diclofenac for the treatment of osteoarthritis pain: a 12 week, phase 3 study. Curr Med Res Opin. 2014 Sep;30(9):1883-93. doi: 10.1185/03007995.2014.946123. Epub 2014 Aug 6. PMID 25050589

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac 35 mg Two Times Daily: Diclofenac (two times daily): Capsules
- Diclofenac 35 mg Three Times Daily: Diclofenac (three times daily): Capsules
- Placebo: Placebo: Capsule
Period: Overall Study
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Started | 104 | 98 | 103
Completed | 91 | 81 | 86
Not Completed | 13 | 17 | 17
Not completed — Lack of Efficacy | 2 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Adverse Event | 9 | 12 | 4
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo | Total
Number analyzed (Participants) | 104 | 98 | 103 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.33) | 61.7 (9.90) | 61.8 (8.42) | 61.6 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 71 | 203
  Male | 40 | 30 | 32 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 8 | 17
  Not Hispanic or Latino | 97 | 96 | 95 | 288
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Subjects were allowed to select more than one race; therefore, some subjects are counted multiple times.
  participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Black or African American | 23 | 14 | 20 | 57
    White or Caucasian | 80 | 83 | 82 | 245
    Other | 0 | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 88.16 (17.037) | 89.35 (16.552) | 89.44 (17.991) | 88.97 (17.167)
Height [Mean (Standard Deviation); unit: cm] | 169.91 (10.561) | 167.60 (9.794) | 168.70 (9.245) | 168.76 (9.898)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (5.18) | 31.8 (5.09) | 31.3 (5.18) | 31.2 (5.16)
Baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score [Mean (Standard Deviation); unit: mm] — The pain in subjects with osteoarthritis was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the mean of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level within the past 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  mm | 73.42 (15.22) | 76.18 (14.15) | 75.27 (17.27) | 74.93 (15.61)
Baseline Total (Composite) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Sc [Mean (Standard Deviation); unit: mm] — The pain, stiffness, and physical function in subjects with osteoarthritis were measured at baseline using the total (composite) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale. The total WOMAC score is the average of the mean visual analogue scale scores, with 0 mm meaning "No Limitation" and 100 mm meaning "Extreme Limitation".
  Baseline total (composite) WOMAC score was calculated for 100 subjects in the Diclofenac Test Capsules two times daily group, 94 subjects in the Diclofenac Test Capsules three times daily group, and 100 subjects in the placebo group.
  mm | 70.26 (15.69) | 72.83 (15.87) | 71.60 (17.24) | 71.54 (16.27)
Baseline Pain Intensity Visual Analogue Scale Score [Mean (Standard Deviation); unit: mm] — The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  The Baseline Pain Intensity VAS score was calculated for 100 subjects in the Diclofenac Test Capsules two times daily group, 94 subjects in the Diclofenac Test Capsules three times daily group, and 100 subjects in the placebo group.
  mm | 69.6 (19.99) | 71.8 (19.33) | 71.5 (18.82) | 71.0 (19.35)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference is calculated as the WOMAC pain subscale score assessed at Week 12 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug and had available measurements at the time specified.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Number analyzed (Participants) | 102 | 96 | 96
mm | -39.04 (2.905) | -44.14 (3.070) | -32.46 (2.937)
Statistical Analysis 1: Comparison: Diclofenac 35 mg Three Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis; Difference in Least Squares Mean = -11.68, 95% CI 2-sided [-19.17 to -4.19], Standard Error of Mean 3.806
Statistical Analysis 2: Comparison: Diclofenac 35 mg Two Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0795, Mixed Models Analysis; Difference in Least Squares Mean = -6.58, 95% CI 2-sided [-13.94 to 0.78], Standard Error of Mean 3.739

2. Secondary Outcome: Change From Baseline to Week 2 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference was calculated as the WOMAC pain subscale score assessed at Week 2 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Number analyzed (Participants) | 100 | 94 | 92
mm | -31.40 (2.742) | -37.42 (2.907) | -21.60 (2.787)
Statistical Analysis 1: Comparison: Diclofenac 35 mg Three Times Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Difference in Least Squares Mean = -15.82, 95% CI 2-sided [-22.82 to -8.83], Standard Error of Mean 3.552
Statistical Analysis 2: Comparison: Diclofenac 35 mg Two Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0052, Mixed Models Analysis; Difference in Least Squares Mean = -9.80, 95% CI 2-sided [-16.66 to -2.95], Standard Error of Mean 3.481

3. Secondary Outcome: Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference was calculated as the WOMAC pain subscale score assessed at Week 6 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Number analyzed (Participants) | 91 | 86 | 87
mm | -36.64 (2.889) | -43.51 (3.051) | -31.08 (2.922)
Statistical Analysis 1: Comparison: Diclofenac 35 mg Three Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Difference in Least Squares Mean = -12.43, 95% CI 2-sided [-19.87 to -4.99], Standard Error of Mean 3.776
Statistical Analysis 2: Comparison: Diclofenac 35 mg Two Times Daily vs Placebo; Test type: Superiority or Other; p = 0.1349, Mixed Models Analysis; Difference in Least Squares Mean = -5.56, 95% CI 2-sided [-12.86 to 1.74], Standard Error of Mean 3.707

4. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference was calculated as the WOMAC pain subscale score assessed at Weeks 2, 6, and 12 minus the average of the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Number analyzed (Participants) | 104 | 98 | 100
mm | -35.62 (2.633) | -41.38 (2.796) | -28.14 (2.647)
Statistical Analysis 1: Comparison: Diclofenac 35 mg Three Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Difference in Least Squares Mean = -13.24, 95% CI 2-sided [-19.89 to -6.59], Standard Error of Mean 3.377
Statistical Analysis 2: Comparison: Diclofenac 35 mg Two Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0248, ANCOVA; Difference in Least Squares Mean = -7.48, 95% CI 2-sided [-14.00 to -0.96], Standard Error of Mean 3.313

5. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Osteoarthritis Pain, Stiffness, and Function Measured Using the Total (Composite) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score.
Description: Pain, stiffness, and function in subjects with osteoarthritis were measured using the Western Ontario and McMaster Universities (WOMAC) Index, which is a 24-item questionnaire. The total (composite) WOMAC score is calculated as the average of the mean visual analogue scale (VAS) scores from the questions in the pain, stiffness, and function subscales. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their response to each of the questions, with 0 mm representing "No Pain, Stiffness, or Difficulty" and 100 mm representing "Extreme Pain, Stiffness, and Difficulty".
  The total (composite) WOMAC score difference was calculated as the total (composite) WOMAC score assessed at Weeks 2, 6, and 12 minus the total (composite) WOMAC score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug and had available measurements at the times specified.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Number analyzed (Participants) | 100 | 94 | 97
mm | -30.25 (2.632) | -35.86 (2.798) | -23.22 (2.656)
Statistical Analysis 1: Comparison: Diclofenac 35 mg Three Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference in Least Squares Mean = -12.63, 95% CI 2-sided [-19.32 to -5.94], Standard Error of Mean 3.396
Statistical Analysis 2: Comparison: Diclofenac 35 mg Two Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0363, ANCOVA; Difference in Least Squares Mean = -7.03, 95% CI 2-sided [-13.60 to -0.45], Standard Error of Mean 3.339

6. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale.
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Pain Imaginable".
  The VAS pain intensity difference is calculated as the average of the VAS pain intensity scores at Weeks 2, 6, and 12 minus the VAS pain intensity at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Number analyzed (Participants) | 104 | 98 | 100
mm | -36.41 (2.670) | -41.33 (2.830) | -30.95 (2.690)
Statistical Analysis 1: Comparison: Diclofenac 35 mg Three Times Daily vs Placebo; Test type: Superiority or Other; p = 0.0028, ANCOVA; Difference in Least Squares Mean = -10.38, 95% CI 2-sided [-17.16 to -3.60], Standard Error of Mean 3.441
Statistical Analysis 2: Comparison: Diclofenac 35 mg Two Times Daily vs Placebo; Test type: Superiority or Other; p = 0.1081, ANCOVA; Difference in Least Squares Mean = -5.46, 95% CI 2-sided [-12.13 to 1.21], Standard Error of Mean 3.385

ADVERSE EVENTS:
Groups:
- Diclofenac 35 mg Two Times Daily: Diclofenac Test (two times daily): Capsules
- Diclofenac 35 mg Three Times Daily: Diclofenac Test (three times daily): Capsules
Arm/Group | Diclofenac 35 mg Two Times Daily | Diclofenac 35 mg Three Times Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 3/104 | 4/98 | 2/103
Other Adverse Events (participants affected / at risk) | 11/104 | 21/98 | 13/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac 35 mg Two Times Daily (N=104) | Diclofenac 35 mg Three Times Daily (N=98) | Placebo (N=103)
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac 35 mg Two Times Daily (N=104) | Diclofenac 35 mg Three Times Daily (N=98) | Placebo (N=103)
Diarrhea (Gastrointestinal disorders) | 5 | 7 | 3
Headache (Nervous system disorders) | 2 | 6 | 3
Nausea (Gastrointestinal disorders) | 5 | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No